CLINICAL TRIAL: NCT00267670
Title: The Effect of Pentoxifylline on Nonalcoholic Steatohepatitis (NASH)
Brief Title: Pentoxifylline/Nonalcoholic Steatohepatitis (NASH) Study: The Effect of Pentoxifylline on NASH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary Rinella, Mary E. Rinella, MD, Northwestern University, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB # 1347-001; GCRC Protocol #891 (Other: Northwestern University Clinical Research Center)
Record Dates: First submitted 2005-12-12; First posted 2005-12-21 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Nonalcoholic Steatohepatitis; Liver Diseases
Keywords: Fatty Liver Disease; Liver; NASH; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease (NAFLD); Pentoxifylline
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — Pentoxifylline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxifylline (Experimental): 400mg PO TID
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): 1 pill PO TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — 400mg PO TID
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — 1 pill PO TID
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the potential benefit of the medication, pentoxifylline, for the treatment of NASH.

DETAILED DESCRIPTION:
This is an investigational study looking at subjects who have been diagnosed with nonalcoholic steatohepatitis (NASH) or 'fatty liver disease'. There is currently no FDA approved available treatment for NASH. The purpose of this study is to explore the potential benefit of the medication, pentoxifylline, for the treatment of NASH. The effectiveness of this drug will be determined by taking blood samples and a liver biopsy. To determine if there is any effect of the medication, two-thirds of the patients participating in the study will receive pentoxifylline and one-third will receive placebo (sugar pill). Thus, an individual's chance of receiving the drug is 67%. In addition to receiving a study drug (placebo or pentoxifylline) the subjects will be encouraged to achieve modest weight loss (~1-2 lbs/week) via low-fat diet and exercise.

The drug (Pentoxifylline) being studied is not approved for use in people who have NASH. Pentoxifylline is considered experimental in this study. Pentoxifylline has been safely used for the treatment of other medical conditions such as alcohol related liver disease and poor circulation. Pentoxifylline is a pill which is taken three times a day.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing to give written informed consent
2. Diagnosis of steatohepatitis Grade >= 1 (Brunt et al. criteria - Am J Gastroenterology 1999;94(9)2467-74) on biopsy within 6 months prior to entry into protocol
3. No histologic evidence of cirrhosis
4. Persistent ALT elevation (> 1.5 the upper limit normal) over 6 months prior to entry into study
5. Adult subjects 18-65 years of age of any race or gender
6. Compensated liver disease with the following hematologic, biochemical, and serological criteria on entry into protocol:

   * Hemoglobin > 11 gm/dL for females and > 12 gm/dL for males
   * White blood cell (WBC) > 2.5 K/UL
   * Neutrophil count > 1.5 K/UL
   * Platelets > 100 K/UL
   * Direct bilirubin, within normal limits
   * Indirect bilirubin within normal limits (unless non-hepatitis factors such as Gilbert's disease explain indirect bilirubin rise. In such cases total bilirubin must be < 3.0 mg/dL)
   * Albumin > 3.2 g/dL
   * Serum creatinine within normal limits
7. Hemoglobin A1c (HgbA1c) < 7%
8. Antinuclear antibodies (ANA) < 1:160
9. Anti-smooth muscle Ab negative
10. Serum hepatitis B surface antigen (HepBsAg) negative
11. Serum hepatitis C antibody (HepC Ab) negative
12. Iron/total iron binding capacity (TIBC) ratio (transferrin saturation) < 45%
13. Alpha-1-antitrypsin level within normal limits
14. Ceruloplasmin level within normal limits
15. Negative pregnancy test (females)
16. Concomitant use of lipid lowering agents at study entry will not exclude patients from the study.

Exclusion Criteria:

1. Evidence of decompensated cirrhosis
2. Active gastrointestinal (GI) bleeding
3. Renal failure (creatinine clearance < 80 mL/min)
4. Active alcohol or drug abuse
5. Uncontrolled diabetes (HgbA1c > 7)
6. Current treatment with anti-diabetic medications such as thiazolidinediones or metformin (stable doses of sulfonylureas are acceptable)
7. Current treatment with anti-TNF alpha medication (i.e. Remicade or Enbrel)
8. Current treatment with vitamin E
9. Alcohol consumption < 20 g/day (males) or < 10 g/day (females) - assessed by one physician and confirmed with one family member.
10. HIV positive status
11. Any history of cerebral and/or retinal hemorrhage
12. Prior intolerance of pentoxifylline or any other methylxanthine (i.e. caffeine, theophylline, or theobromine)
13. Current use of theophylline
14. Known diagnosis of malignancy
15. Any other conditions which the investigator feels would make the subject unsuitable for enrollment, or could interfere with the subject completing the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Rinella, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Van Wagner LB, Koppe SW, Brunt EM, Gottstein J, Gardikiotes K, Green RM, Rinella ME. Pentoxifylline for the treatment of non-alcoholic steatohepatitis: a randomized controlled trial. Ann Hepatol. 2011 Jul-Sep;10(3):277-86. PMID 21677329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2005 to March 2008 patients were recruited through the Northwestern Memorial Faculty Foundation Hepatology Clinic.
Pre-assignment Details: Subjects were excluded from the study if they had evidence of another form of liver disease or if they were HIV positive, pregnant or had evidence of ongoing alcohol consumption exceeding 20g(males) and 10g(females)daily. Furthermore, subjects were excluded if they were taking drugs known to cause steatohepatitis.
Groups:
- Pentoxifylline: This group was given pentoxifylline 400mg thrice daily (tid) for 1 year
- Placebo: This group was given a capsule identical to pentoxifylline that contained sucrose.
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 19 | 7
Completed | 15 | 7
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pentoxifylline: Patients in this group received pentoxifylline 400mg tid for 1 year.
- Placebo: Patients in this group received a capsule identical to pentoxifylline that instead contained sucrose.
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 19 | 7 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 7 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10) | 53 (8) | 49.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 19 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a 30% Reduction in Alanine Aminotransferase (ALT) Treated With Pentoxifylline (PTX) or Placebo for 12 Months.
Description: The primary goal of the study was to determine whether pentoxifylline (PTX) therapy improved serum ALT (> or = 30% change from baseline to month 12) compared to placebo.
Time Frame: baseline and 12 months
Population: The primary analysis was done as intention to treat. A secondary analysis was performed per protocol and there were no differences between the two analyses. Intention to treat results are reported.
Measure: Number; unit: participants
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 19 | 7
participants | 19 | 7
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Sample size estimates were based on 30% reduction in ALT in the treatment group & 15% reduction in the placebo group. With a sample size of 30 planned (20 treatment:10 placebo), the study was designed to have a power of 90% to detect a difference in means of 1.25 standard deviations (ES=1.25), & a power of 80% to detect a difference in means of 1.1 standard deviations (ES=1.1), based on calculations using power index, z-table, & accounting for unequal sample size: n1 = 20, n2 = 10, a = 0.05; Test type: Superiority or Other; p = 0.46, ANOVA; Odds Ratio (OR) = 1, Standard Error of Mean 1

2. Secondary Outcome: The Effect of Pentoxifylline on Change in Tumor Necrosis Factor [TNF]-α Levels in Patients With NASH
Description: The mean change from baseline to month 12 in proinflammatory cytokines (such as TNF-α) and gene expresssion were the secondary endpoints and were analyzed with the same analysis of covariance model and summary statistics specified for the primary endpoint. Differences were regarded as statistically significant when P < 0.05. The results for TNF-α are reported here. Interleukin-6 [IL-6], IL-10) and expression of TNF-alpha Receptors (p55 and p75) had insufficient data for statistical analysis.
Time Frame: one year
Population: Intention to Treat with last observation carried forward
Measure: Mean (Standard Error); unit: pg/dL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 19 | 7
pg/dL | -117.9 (109.5) | 18.3 (64.4)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Null hypothesis was that there was no difference between mean hepatic expression of TNF-alpha receptors in patient with NASH. This was a secondary outcome and no power analysis was done; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

3. Secondary Outcome: Change in Serum Leptin Levels in Patients Treated With Pentoxifylline or Placebo for 12 Months
Description: Values represent changes in leptin from baseline to 12 months in patients treated with pentoxifylline or placebo.
Time Frame: baseline and one year
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Placebo: Patients in this group received a capsule identical to pentoxifylline that instead contained sucrose thrice daily for 1 year.
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 19 | 7
ng/mL | 0.78 (0.07) | 0.78 (0.08)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Test type: Superiority or Other; p = 0.94, t-test, 2 sided

4. Secondary Outcome: Change in Serum Adiponectin Levels in Patients Treated With Pentoxifylline or Placebo for 12 Months
Time Frame: one year
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 19 | 7
ug/mL | 0.4 (0.3) | 0.8 (0.4)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 1 year for the duration of the study.
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/7
Other Adverse Events (participants affected / at risk) | 0/19 | 0/7

LIMITATIONS AND CAVEATS:
The most significant limitation of this study is the small sample size, thus the lack of statistical significance may be due to low power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes